CLINICAL TRIAL: NCT04052230
Title: Evolution of Diaphragm Thickness Under Veno-arterial ECMO : Observational Study
Brief Title: Evolution of Diaphragm Thickness Under Veno-arterial ECMO
Acronym: ATROPHY-ECMO
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.142; 2019-A01273-54 (Other: ID RCB)
Record Dates: First submitted 2019-06-11; First posted 2019-08-09 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Diaphragm; Extracorporeal Membrane Oxygenation Complication
Keywords: diaphragm; ECMO; ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ultrasound measure — Admission to the intensive care unit, and setting up an ECMO Daily monitoring from D1 to D7, follow up at D60

SUMMARY:
The main objective is to evaluate the evolution of the thickness of the diaphragm (during the first week of treatment) by VA ECMO in the resuscitation patients.

The comprehension of the mechanisms involved in the diaphragm ailment will identify modifiable factors that lead to muscle degradation and thus to the deterioration of patients' prognosis.

DETAILED DESCRIPTION:
The evolution of diaphragm muscle thickness is described in human resuscitation under mechanical ventilation, but the incidence, causes and functional impact have not been studied in patients undergoing cardiopulmonary bypass ECMO (extra-corporeal membrane oxygenation) veno-arterial (VA). More generally, the muscular mechanisms of dyspnea in cases of acute cardiac dysfunction are not known.

The evolution of the diaphragmatic thickness in intensive care has been described during prolonged stay in intensive care and from the initial phase of septic status. It is associated with dyspnea, weaning delay of mechanical ventilation and impact on patient outcomes. The atrophy of the diaphragm muscle is related to both loss of function and loss of muscle performance. The same is true for hypertrophy that is caused by overuse of the muscle and also causes loss of function.

Decreased cardiac muscle performance may require both cardiac assistance and respiratory assistance. Cardiac and respiratory dysfunction may complicate withdrawal of respiratory assistance and extracorporeal circulatory support devices. These two supports, respiratory and circulatory support, make it possible to mitigate the insufficiency of the systemic flow, the oxygenation and the purification of the CO2. Respiratory assistance is known to influence the diaphragmatic function. The role of muscle pump function in the weaning process of the ECMO, however, remains largely unknown.

Ultrasound is used in the patient's bed in daily practice to measure cardiac function, the study of vessels but also the diaphragm muscle. It allows to study the trophicity of the diaphragm and these efforts via its contraction. The hypothesis that there is muscular involvement of the diaphragm in this measurable condition by ultrasound method can be formulated.

No study has systematically explored the existence of diaphragmatic atrophy under VA ECMO. The influence of cardiac and respiratory assistance is not known.

The purpose of this study is to provide a description of the diaphragm physiology of patients treated with VA ECMO.

It is to evaluate the evolution of the trophicity of the diaphragm muscle in intensive care.

Secondly, to evaluate the factors that influence it at the time of weaning. In this study it's planed to include a cohort of patients with a longitudinal evaluation of the thickness of the diaphragm during a cardiogenic shock under ECMO, and an evaluation of the influence of ECMO parameters and ventilation on the diaphragm.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in intensive care
* Patient under veno-arterial ECMO
* Non-opposition of the patient or relatives
* Affiliation to a health insurance

Exclusion Criteria:

* Subject under guardianship or subject deprived of liberty
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is adult patients hospitalized in intensive care for circulatory insufficiency requiring assistance with ECMO VA.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-10-13 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
To evaluate the evolution of the trophicity of the diaphragm muscle during the first week of treatment with VA ECMO in patients in intensive care. | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Evaluation of the trophicity of the diaphragm muscle at the end of the expiration from the first day in the intensive care unit after the ECMO implementation until the D7 of the hospitalization with ultrasound. A change greater than 10% of the thickness will define three groups of patients (loss of thickness, stability and thickness gain). The first day that this value is reached will determine the allocation in one or the other group.

SECONDARY OUTCOMES:
To evaluate the evolution of the performance of the diaphragm muscle in patients in intensive care. | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the thickening fraction of the diaphragm.
To evaluate the link between the evolution of respiratory physiological variables and the diaphragm evolution in patients in intensive care. | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily evolution of tidal volume during ultrasound collection
To evaluate the link between the evolution of respiratory physiological variables and the diaphragm evolution in patients in intensive care. | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily evolution of respiratory rate during ultrasound collection
To evaluate the link between the evolution of respiratory physiological variables and the diaphragm evolution in patients in intensive care. | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily evolution of pulse oximetry during ultrasound collection
To evaluate the link between the evolution of respiratory physiological variables and the diaphragm evolution in patients in intensive care. | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily evolution of occlusion pressure at 100ms (P0.1)during ultrasound collection
To evaluate the link between the evolution of respiratory physiological variables and the diaphragm evolution in patients in intensive care. | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily evolution of maximum inspiratory pressure (MIP) during ultrasound collection
To evaluate the link between the evolution of respiratory physiological variables and the diaphragm evolution in patients in intensive care. | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily evolution of SNIFF test during ultrasound collection
To evaluate the link between parameters of mechanical ventilation and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily ventilatory mode
To evaluate the link between parameters of mechanical ventilation and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily tidal volume
To evaluate the link between parameters of mechanical ventilation and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily respiratory rate
To evaluate the link between parameters of mechanical ventilation and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily positive expiratory pressure
To evaluate the link between parameters of mechanical ventilation and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily plateau pressure
To evaluate the link between parameters of mechanical ventilation and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily motor pressure
To evaluate the link between parameters of mechanical ventilation and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily transpulmonary pressure
To evaluate the link between parameters of mechanical ventilation and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily oesophageal pressure
To evaluate the link between parameters of mechanical ventilation and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily O2 inspired fraction.
To evaluate the link between the impact of ECMO parameters and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily the daily blood flow
To evaluate the link between the impact of ECMO parameters and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily the daily sweep rate
To evaluate the link between the impact of ECMO parameters and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily the daily oxygenation
To evaluate the link between the impact of ECMO parameters and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily percentage of the theoretical flow
To evaluate the link between the impact of ECMO parameters and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily duration of ECMO
To evaluate the link between the impact of ECMO parameters and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  Measurement of the daily the success of weaning.
To evaluate the link between the associated organ failures and the diaphragm evolution in patients in intensive care | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, and Day 7
  The daily change in the incidence of diaphragmatic dysfunction defined by the diaphragm thickening fraction <20% during a maximal inspiratory test to J7. The daily collection of hemodynamic variables during the diaphragmatic ultrasound collection including an evaluation of the visual LVEF.
To evaluate the impact of the diaphragm evolution on the future of the patient in intensive care: weaning of the assistances, survivals.and the diaphragm | Day 60
  Measurement of the survival
To evaluate the impact of the diaphragm evolution on the future of the patient in intensive care: weaning of the assistances, survivals.and the diaphragm | Day 60
  Measurement of the length of stay in intensive care unit
To evaluate the impact of the diaphragm evolution on the future of the patient in intensive care: weaning of the assistances, survivals.and the diaphragm | Day 60
  Measurement of the failure of extubation
To evaluate the impact of the diaphragm evolution on the future of the patient in intensive care: weaning of the assistances, survivals.and the diaphragm | Day 60
  Measurement of the number of days without mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France